CLINICAL TRIAL: NCT03642093
Title: H.O.P.E. Healing Optimization Through Preoperative Engagement: A Prospective Single Cohort Study to Evaluate the Effect of a Prehabilitation Program on Preoperative Outcomes in Upper GI Surgical Oncology Patients
Brief Title: HOPE - A Study to Evaluate the Effect of a Prehabilitation Program on GI Cancer Patients Planning to Undergo Surgery
Acronym: HOPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Siobhan Trotter (Other)
Responsible Party: Sponsor-Investigator, Siobhan Trotter, Nurse Practitioner, Preoperative Optimization Program, Surgical Oncology and General Surgery, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOPE Study 2018.045
Record Dates: First submitted 2018-06-20; First posted 2018-08-22 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Cancer; Esophageal Cancer; Gastric Cancer
Keywords: Frailty; Prehabilitation
MeSH Terms: conditions — Pancreatic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Frailty | interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Frail (Experimental): Subjects assessed and determined to be Frail and meet trial eligibility criteria will be enrolled on Frail Arm and begin a 4 Week program consisting of Nutritional Interventions and Physical Activity Interventions
  Interventions: Combination Product: Nutritional Intervention; Behavioral: Physical Activity Intervention
- Not Frail (Active Comparator): Subjects assessed and determined to be Not Frail and meet trial eligibility criteria will be enrolled on Not Frail Arm and begin a 4 Week program consisting of Nutritional Interventions and Physical Activity Interventions
  Interventions: Combination Product: Nutritional Intervention; Behavioral: Physical Activity Intervention

INTERVENTIONS:
Combination Product: Nutritional Intervention — Nutritional Supplementation for all subjects and Pancreatic Enzyme Replacement Therapy only for subjects with Exocrine Pancreatic Insufficiency
  Other Names: Immunonutrition
Behavioral: Physical Activity Intervention — Walking and Inspiratory Muscle Training

SUMMARY:
A one-group prospective cohort study design with measures collected pre- and post-intervention. The primary goal of this study is to evaluate the effect of a multimodal prehabilitation preoperative program on changes in frailty in upper gastrointestinal surgical oncology patients.

DETAILED DESCRIPTION:
Cancer patients often develop protein calorie malnutrition, inflammatory states, and loss of lean muscle mass, which can be best categorized as frailty. Frailty affects global health, the ability to carry out normal functions, and even the ability to tolerate targeted curative treatments such as surgery, chemotherapy, and radiation. The Investigators evaluate frailty, and design a study to evaluate the outcomes of the administration of multimodal preoperative prehabilitation programs on those frailty markers. Previous data provides support for interventions that include:

1. Improved protein rich nutrition with specific immunonutrition recommendations,
2. Treatment of maldigestion or pancreatic insufficiency in pancreatic, gastric, or esophageal cancer patients,
3. Brief, evidence-based activity interventions such as walking and inspiratory muscle training (IMT), and
4. Disease specific education

These interventions should improve frailty by maintaining or regaining weight, improved grip strength, and improved prealbumin. These markers indicate improvements in nutritional status, increased strength and ability to ambulate, and improved functional status in the preoperative period. Other outcomes that will be reported include fat-soluble vitamin levels, global health, and inflammation.

The preoperative period is the best time to facilitate patient engagement through self-care and proactive activity. Interventions must be easy to accomplish and structured so patients have accountability and both patients and clinicians have methods and tools for measuring progress. Most patients and family members are motivated at this time and understand the need to improve frailty and potentially improve global health.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be patients of Ochsner being seen at the Ochsner Medical Center (OMC).
* All patients must be 25 to 80 years of age.
* All patients must have a diagnosis of cancer.
* > 10 pound unintentional weight loss within 1 year
* Ability to perform grip strength test and Timed Up and Go (TUG) test
* Willingness to participate in the study, document compliance, and attend clinical appointments
* All patients must be undergoing one of the following major elective surgical oncologic resections with curative intent:

  * Pancreaticoduodenectomy for pancreatic cancer
  * Distal pancreatectomy / splenectomy for pancreatic cancer
  * Esophageal robotic assisted laparoscopic thoracoscopic esophagectomy for esophageal cancer
  * Laparoscopic or open, partial or total gastrectomy for gastric cancer

Exclusion Criteria:

* All patients not undergoing oncologic or major resections.
* All patients unwilling or unable to answer questionnaires or accept help to answer electronic or paper questionnaires.
* All patients that are unable to participate in an activity program.
* All patients unable to wear an electronic activity monitoring device.
* All patients not wanting to follow a specific nutritional and breathing intervention.
* All patients that are not able or wishing to consent.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Frailty Measurement | 4 Weeks
  Frailty will be measured using 3 criteria: weight loss, grip strength, and prealbumin serum level

SECONDARY OUTCOMES:
Vitamin levels | 4 Weeks
Quality of Life (QoL) Assessment | 4 Weeks
  QoL will be assessed using Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Questionnaire - PROMIS Scale v1.2 - Global Health

CONTACTS AND LOCATIONS:
Overall Officials: Siobhan M Trotter, DNP, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Medical Center, New Orleans, Louisiana, United States